CLINICAL TRIAL: NCT04516473
Title: The Impact of Abdominal Body Contouring Surgery on Physical Function After a Massive Weight Loss: a Non-randomized Control Trial
Brief Title: The Impact of Abdominal Body Contouring Surgery on Physical Function After a Massive Weight Loss (BCSP)
Acronym: BCSP
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Cameron Mitchell, Assistant Professor, University of British Columbia
Other Study IDs: H20-00960
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Weight Loss; Obesity
Keywords: Panniculectomy; Excess Skin
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental/Body Contouring Intervention: These are participants who have self-selected to undergo an abdominal body contouring procedure within the course of the study.
  Interventions: Procedure: Abdominal Body Contouring
- Control/Post Massive Weight Loss Matched Control: These are participants who have similar characteristics to the body contouring intervention group, but they will not undergo any surgical procedure during the course of the study.
  The addition of this matched control group with a similar degree of excess skin but who will not be undergoing body contouring surgery will control for any changes in physical function which may occur without any intervention within the testing sessions. This group will also control for any learning effects between testing sessions.

INTERVENTIONS:
Procedure: Abdominal Body Contouring — These are surgeries that correct for excess skin and its adverse consequences. The surgeries that focus on central area to remove a large hanging pannus is usually called panniculectomies or abdominoplasties; the former is focused on the excision of excess tissue to relieve impairment while the latter is generally considered a cosmetic surgery. The form of the surgery is case dependent and can range from removing apron of skin to complete contouring of the abdomen with tightening of the abdominal muscle and moving the belly button.
  Groups: Experimental/Body Contouring Intervention

SUMMARY:
Obesity is a growing chronic medical condition in which as of 2015, a total of 107.7 million children and 603.7 million adults were considered obese and since 1980 the prevalence of obesity has doubled in more than 70 countries. It is estimated that 70 percent of individuals who undergo a massive weight loss would develop excess skin and based on patient reported outcome measures, it has been shown that excess skin negatively impacts patients' body image, self-esteem, physical function and body contouring surgeries have been demonstrated to improve these measures. These are surgeries that correct for excess skin and its adverse consequences. The form of the surgery is case dependent and can range from removing an apron of skin to complete contouring of the abdomen with tightening of the abdominal muscle and moving the belly button. Despite previous studies indicating mobility limitation because of excess skin and improvements after abdominal body contouring surgeries with the use of subjective measures of physical function, there are no studies that directly measures physical fitness post body contouring surgeries. Therefore, the purpose of the current study is to evaluate the impact of abdominal body contouring surgeries on direct objective measures of physical function.

It is hypothesized that 1) the removal of excess skin will improve direct objective measures of physical function in post massive weight loss participants 2) the removal of excess skin will improve direct measures of gait and balance in post massive weight loss participants 3) the removal of excess skin will improve patient reported outcome measures using quality of life questionnaires in post massive weight loss participants 4) the removal of excess skin will improve aerobic capacity in post massive weight loss participants 5) the removal of excess skin does not change the body composition in post massive weight loss participants.

DETAILED DESCRIPTION:
Participants will be recruited through multiple medical clinics and will visit the exercise, nutrition and muscle metabolism lab twice over the course of 8-12 weeks to complete objective and subjective measures of physical function. Each testing session will be conducted by the study investigator and physical function testing will be video recorded to reduce measurer bias. Based on participants' status they will be allocated to either a body contouring intervention group (BCI) or a post massive weight loss matched control (PMWMC). The first testing session would happen preoperatively and second one would happen between 8-12 weeks postoperatively depending on recovery required. Pain levels will be measured both pre and postoperatively using a numerical rating scale (0-10) to ensure adequate recovery.

Outcomes will include a variety of objective measures of physical function including 9-item modified physical performance test (mPPT), 30 second chair stand, timed up and go, stair climbing power, modified agility t-test, star excursion balance test, and 6 minute walk test. A body composition measure consisting of fat mass and fat free mass will also be obtained via dual-energy X-ray absorptiometry. Subjective measures would include 6 components of health related quality of life measure using BODY-Q questionnaire that would include sub scales such as body image, physical function, psychological, sexual, social, and obesity symptoms. Other subjective measure would include rate of perceived exertion which would be measured during each of the objective tests.

Additionally, grade of excess skin would be measured by images provided to the participants and weight of the resected excess skin will be obtained from the operating surgeon at the end of the study.

To obtain demographic history, physical activity level post surgery and to gain feedback for future clinical trial, the participants will also complete a socioeconomic status questionnaire, physical activity questionnaire, and participant experience with research questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Weight has not deviated by greater than 5 percent for 3 months
* Have excess grade skin of greater or equal to 2
* Percent total weight loss pre-body contouring of greater or equal to 25 percent
* Fluently read and write English

Exclusion Criteria:

* Any musculoskeletal issues that would prevent participants from doing the physical function tests.
* Current medication history indicating atypical antipsychotics including but not limited to clozapine, olanzapine, quetiapine, risperidone, aripiprazole, amisulpride, ziprasidone, asenapine, iloperidone, lurasidone and paliperidone.
* Severe pulmonary conditions such as severe chronic obstructive pulmonary disease (COPD) and or severe asthma.
* Participants who actively aiming to lose weight
* Have diabetes with diabetic neuropathy or experienced hypoglycemic event within 6 months prior to the study
* Severe kidney disease with estimated glomerular filtration rate (eGFR) less than 60 ml/min
* Pregnant individuals
* Uncontrolled hypertension with resting blood pressure greater than 160/90 mmHg
* Uncontrolled obstructive sleep apnea with symptoms
* On statin therapy with myopathy
* Unstable atrial fibrillation
* Weight pre-body contouring greater than 340 lbs (154 kg)
* Current smoker

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and female who have undergone a massive weight loss through any weight loss intervention, have excess skin, are healthy enough to perform simple physical function tasks and self-selected to undergo abdominal skin removal surgery.
  Participants who have similar criteria to the intervention group but will not undergo surgical intervention during the course of the study will serve as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Change in physical function aggregate score | 8-12 weeks
  Measured by 9-item modified physical performance test that gives an aggregate score out 36 and comprises of 9 tests pre and post surgery and includes the following:
  1. Time to complete a book lift
  2. Time to complete putting on/off a lab coat
  3. Time to complete picking up a penny from the floor
  4. Time to complete a 5 times chair stand
  5. Turning 360 degrees
  6. Time to complete a 50 feet walk
  7. Time to complete 1 flight of stairs
  8. Completing 4 flights of stairs
  9. A progressive romberg test
  Lowest score is 0, highest score is 36 and higher scores represent better outcomes.

SECONDARY OUTCOMES:
Change in lower body strength | 8-12 weeks
  Measured by number of stands completed during a 30 seconds chair stand pre and post surgery
Change in time to complete agility drill | 8-12 weeks
  Measured by time to complete a modified agility t-test pre and post surgery
Change in timed up and go | 8-12 weeks
  Measured by time to complete a timed up and go test
Change in stair climbing power | 8-12 weeks
  Measured by time to ascend 10 stairs and deriving power pre and post surgery
Change in dynamic balance balance | 8-12 weeks
  Measured by star excursion balance test pre and post surgery
Change in aerobic capacity | 8-12 weeks
  Measured by distance traveled during a 6 minute walk test pre and post surgery
Change in lean body mass | 8-12 weeks
  Measured by change in bone free fat mass by using dual-energy X-ray absorptiometry pre and post surgery
Change in fat mass | 8-12 weeks
  Measured by using dual-energy X-ray absorptiometry pre and post surgery
Change in patient reported outcome measure of physical function and quality of life | 8-12 weeks
  Measured by 6 health related quality of life components of BODY-Q questionnaire pre and post surgery. Sub-scales would include body image, physical function, psychological, sexual, social, and obesity/physical symptoms. Each sub-scale will be graded individually, and the raw scores will be converted into a score from 0-100. For body image, physical function, psychological function, sexual, and social function higher scores represent a better outcome
  For obesity/physical symptoms, symptoms will be added so that the total number of symptoms experienced would be obtained. Minimum number of symptoms is 0 and maximum is 10.
Change in rate of perceived exertion (RPE) during physical function tests | 8-12 weeks
  Measured by BORG RPE scale pre and post surgery. Minimum score is 6 and maximum is 20. The scale is only to provide how much the participants are being exerted when given a task.

OTHER OUTCOMES:
Correlation between degree of excess skin and change in objective physical function test scores | 8-12 weeks
  Measured by linear models and correlating the degree of excess skin and change in measures of physical function scores from post to pre surgery
Correlation between the weight of resected excess skin and change in objective physical function tests | 8-12 weeks
  Measured by linear models and correlating the amount of weight of the resected excess skin and change in measures of physical function scores from post to pre surgery

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Mitchell, PhD, Principal Investigator — Assistant Professor University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
No plan available for IPD sharing